Study: Health Opportunities & Promoters of Equitable Screening for Lung Cancer (HOPES for

Lung Cancer) 1K08CA270430-01A1

Date of Approval: 1.17.23

Principal Investigator: Efren J. Flores, MD

Contact:

**Phone:** 617-643-9420

Email: ejflores@mgh.harvard.edu OR arlin arias@dfci.harvard.edu

**Purpose of the Research**: The goal of this study is to reduce Lung Cancer Screening (LCS) disparities among the Latino/Hispanic community by addressing issues and obstacles that patients, patient advocates, providers and medical systems face. LCS can help detect lung cancer early, which can increase the chance of effective treatment. Understanding how we can and improving how we currently document smoking history and patient status will help improve existing outreach and patient care, reducing the existing barriers that negatively impact the community.

**Study Information**: You are being asked to participate in a focus group with other patients and patient advocates because we think you will provide helpful feedback about improving smoking history documentation and the development of an educational video. We will use a series of open-ended questions to guide the discussion in which we will discuss patients' reasons for smoking disclosure and barriers to lung cancer screening. The information you share in the group session will guide us in refining best practices to improve smoking history documentation in electronic health records system (EHR) and outreach methods.

This focus group discussion will be an opportunity to have an open dialogue where there are no right or wrong answers. We are not aiming to reach a consensus on anything. Your honest answers and ideas will be instrumental in our process of improving EHR. I am interested in hearing all of your thoughts and ideas. If you do not want to answer a particular question, you are not obligated to answer as participation is voluntary.

**Time Required:** 1 hour over two days

**Risks and Benefits:** The benefit of your participation is that you may better understand the benefits of lung cancer screening, and you will help inform our outreach.

**Compensation:** After you participate in the group session and fill out the questionnaire, we will give you a \$30 gift card in appreciation of your time. If you participate in the follow-up survey about the educational outreach, we will provide an additional \$5.

Confidentiality: We will audio record the focus group conversation in order to remember and professionally transcribe anonymously the content that has been shared. Your participation involves little risk because all the information transcribed and submitted will be anonymous. All audio recordings will be deleted once the transcription process is complete. The only people who will read this transcript will be our trained research staff. If we use the information you share, such as for publication, presentation at a meeting, or a future training program, we will ensure complete confidentiality of your responses.

The focus group discussion will be strictly confidential. By keeping what is said in the focus group private, we can discuss our experiences comfortably as a group. This will allow us to preserve the safety and privacy for each of you to speak openly. We will be extremely careful to protect your privacy by locking all study materials in file cabinets and storing data on password-protected computers to which only our study team has access. While researchers can never guarantee complete confidentiality of study data, I assure you that we will take all efforts to prioritize data security. If the results of this research study are published in a medical journal, they will not identify individual participants.

**Voluntary Participation:** Your participation in this study is completely voluntary. There is no penalty for not participating, and you do not have to answer any question you do not wish to answer.

**Right to withdraw from the study:** You have the right to withdraw from the study at any time without consequence. Deciding not to participate won't affect medical care you receive at Mass General Brigham now or in the future, or any benefits they receive now or have a right to receive.

If you'd like to speak to someone not involved in this research about your rights as a research subject, or any concerns or complaints you may have about the research, contact the Mass General Brigham IRB at (857) 282-1900.

We are required by the Health Insurance Portability and Accountability Act (HIPAA) to protect the privacy of health information obtained for research. This is an abbreviated notice, and does not describe all details of this requirement. During this study, identifiable information about you or your health will be collected and shared with the researchers conducting the research. In general, under federal law, identifiable health information is private. However, there are exceptions to this rule. In some cases, others may see your identifiable health information for purposes of research oversight, quality control, public health and safety, or law enforcement. We share your health information only when we must, and we ask anyone who receives it from us to protect your privacy.